CLINICAL TRIAL: NCT02339324
Title: Neoadjuvant Combination Biotherapy With Pembrolizumab and High Dose IFN-alfa2b in Patients With Locally/Regionally Advanced/Recurrent Melanoma: Safety, Efficacy and Biomarker Study
Brief Title: Neoadjuvant Combination Biotherapy With Pembrolizumab and High Dose IFN-alfa2b
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yana Najjar (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Yana Najjar, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCI 14-102
Record Dates: First submitted 2014-12-07; First posted 2015-01-15 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Interferon alpha-2; Introns

STUDY DESIGN:
Intervention Model Description: PI will be leaving this institution and has elected to close this trial to accrual
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- This study has one arm that consists of 3 phases or steps. (Experimental): Induction phase (first 6 weeks): Pembrolizumab and High Dose IFNα-2b (HDI) Pembrolizumab I.V. every 3-4 weeks for 2 doses concurrently with HDI I.V. x 5 consecutive days every week for 4 weeks, followed by S.C. every other day 3x each week for 2 weeks.
  Surgery phase (week 6-8).
  Maintenance phase (following recovery from surgery): Pembrolizumab I.V. infusion every 3 weeks given concurrently with HDI S.C. QOD (e.g. M,W,F) TIW every week for 46 additional weeks
  Interventions: Drug: Pembrolizumab and high dose interferon alfa-2b (HDI)

INTERVENTIONS:
Drug: Pembrolizumab and high dose interferon alfa-2b (HDI) — Pembrolizumab and HDI will be given concurrently during the induction phase of the study for up to 6 weeks from treatment initiation. This is followed by surgery. After recovery from surgery, pembrolizumab and HDI will be reinitiated as maintenance therapy during the maintenance phase of the study.
  Other Names: MK-3475 and Intron A

SUMMARY:
This study plans to to estimate the safety profile of the combination biotherapy regimen consisting of standard-dose interferon alpha-2b (HDI) and anti-PD1 monoclonal antibody, Pembrolizumab, for the neoadjuvant therapy of locally/regionally advanced/recurrent melanoma. Also, the objectives of this trial include the evaluation of prognostic and predictive biomarkers, radiologic preoperative response rate, pathologic response rate, progression free survival and overall survival. Up to 30 evaluable patients will be accrued.

DETAILED DESCRIPTION:
The study has 3 main phases:

Induction Phase:

Pembrolizumab I.V. infusion every 3-4 weeks for 2 doses (starting first week of HDI administration) given concurrently with HDI I.V. x 5 consecutive days out of 7 every week for 4 weeks, followed by S.C. every other day 3 times each week for 2 weeks.

This is followed by definitive surgery (week 6-8).

Maintenance Phase (following recovery from surgery):

Pembrolizumab I.V. infusion every 3 weeks given concurrently with HDI S.C. QOD TIW every week for 46 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent.
2. At least 18 years of age.
3. Melanoma belonging to the following stages:

   * Tx or T1-4 and
   * N1b, or N2b, or N2c, or N3 and
   * M 0

   Pts are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal and/or in-transit metastasis, or at the time of clinically detected nodal and/or in-transit recurrence and may belong to any of the following groups:
   * Primary melanoma with clinically apparent regional lymph node metastases.
   * Clinically detected recurrence of melanoma at the proximal regional lymph node(s) basin.
   * Clinically detected primary melanoma involving multiple regional nodal groups.
   * Clinically detected single site of nodal metastatic melanoma arising from an unknown primary.
   * Pts with intransit or satelite metastases with or without lymph node involvement are allowed if they are considered potentially surgically resectable at baseline.

   NOTE: A pt should be determined to be potentially surgically resectable at baseline to be eligible for this neoadjuvant study.
4. Have measurable disease.
5. Provide tumor tissue from a newly obtained biopsy.
6. ECOG performance status of 0 or 1.
7. Adequate organ function.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 wks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 wks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
5. Has an active automimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
6. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
7. Has an active infection requiring systemic therapy.
8. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
9. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
10. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
11. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways). Prior treatment with interferon alfa is allowed. Patients with history of allergic or hypersensitivity reaction to interferon alfa are excluded.
12. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
13. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
14. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
The number of participants who experience adverse events. | Up to 90 days (per patient); Up to 5 years (for cohort)

SECONDARY OUTCOMES:
Evaluate changes in immunologic biomarkers in the blood and in the tumor tissue and assess their association with resposne to treatment. | Up to 5 years

OTHER OUTCOMES:
radiologic preoperative response rate | Up to 5 years
pathologic response rate | Up to 5 years
progression free survival | Up to 5 years
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yana Najjar, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No